CLINICAL TRIAL: NCT01134510
Title: A Phase I/II Trial to Evaluate the Safety & Tolerability of Berinert® (C1 Inhibitor) Therapy to Prevent Complement-Dependent, Antibody-Mediated Rejection Post-Transplant in Highly-HLA Sensitized Patients"
Brief Title: Safety & Tolerability of Berinert® (C1 Inhibitor) Therapy to Prevent Rejection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanley Jordan, MD (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor-Investigator, Stanley Jordan, MD, Medical Director, Medical Director, Renal Transplantation & Transplant Immunotherpay, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C1INH001CSMC
Record Dates: First submitted 2010-05-26; First posted 2010-06-02 (Estimated); Results first posted 2015-08-03 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Kidney Transplantation
Keywords: Kidney transplantation
MeSH Terms: interventions — Complement C1 Inhibitor Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- C1 esterase inhibitor (Experimental): 10 subjects will receive C1 esterase inhibitor in addition to standard of care immunosuppressive therapy.
  Interventions: Drug: C1 Esterase Inhibitor
- Placebo (Placebo Comparator): 10 subjects placebo [normal saline] in addition to standard of care immunosuppressive therapy.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: C1 Esterase Inhibitor — C1 Esterase Inhibitor 20 units/kg twice weekly x 4 weeks
  Other Names: Berinert
  Arms: C1 esterase inhibitor
Drug: Placebos — NS (comparable volume as intervention) twice weekly x 4wks
  Arms: Placebo

SUMMARY:
Organ transplantation offers the only hope for a normal life for patients with end-stage renal disease on dialysis (ESRD). For the highly-sensitized patient, patients with antibodies to human leukocyte antigens (HLA), transplantation is extremely difficult or impossible since pre-formed antibodies will cause severe rejection and loss of transplanted organs. Approximately 30% of the transplant list in the U.S. is considered sensitized (have detectable antibodies to HLA antigens). These anti-HLA (anti-Human Leukocyte Antigen antibodies) pose a significant barrier to transplantation that has recently been successfully addressed using desensitization therapies with IVIG, rituximab and/or plasmapheresis (PE). Despite the success of these therapies, post-transplant antibody mediated rejection (AMR) and chronic Antibody Mediated Rejection (CAMR) remain significant problems. Recent data suggests that addition of Berinert (C1 Inhibitor) to post-transplant treatment regimen may significantly reduce incidence of Antibody Mediation Rejection.

Twenty highly-sensitized patients who have undergone desensitization treatment and are awaiting kidney transplant will be enrolled in the study. Once transplanted these patients will be started on the standard of care post-transplant immunosuppressive protocol. In addition patients will receive Berinert 20 units/ kg daily x 3 days, then twice weekly x 3 weeks. At the end of Berinert treatment a kidney biopsy will be performed. Subjects will be followed for 6 months to assess safety and efficacy of the study protocol.

DETAILED DESCRIPTION:
Single center, Phase I/II, randomized The trial will examine the safety and efficacy of human C1 INH given post-transplant to reduce or prevent complement-dependent, antibody-mediated rejection (AMR) in 20 subjects (adult) who are highly-HLA sensitized (HS),(Panel Reactive Antibodies >30% (PRA), have undergone desensitization with intravenous immunoglobin (IVIG) + rituximab and/or plasmapheresis and are awaiting Living donor (LD)/ Deceased Donor (DD) kidney transplant. Once transplant offers are entertained, a donor-specific crossmatch will be performed to detect anti-HLA antibodies and donor-specific anti-HLA antibodies (DSA) which are associated with acute rejection or graft loss. (These anti-HLA (anti-Human Leukocyte Antigen antibodies) antibodies may result naturally or from previous pregnancy, transfusions, or prior transplants.) If acceptable crossmatches and Donor Specific Antibody levels are seen after desensitization, the patients will proceed to Living Donor/Deceased Donor transplantation. Patients receiving transplants will have pre-transplant labs obtained for C1 INH levels, Complement 3 (C3) and Complement 4 (C4) at transplant. In addition to the standard post-transplant immunosuppressive protocol, participating patients will receive placebo or 20 Units/kg C1 INH twice weekly X 4 weeks. At the end of the treatment, a protocol biopsy will be performed to assess the allograft for evidence of Antibody Mediated Rejection, including C4d staining. Since ~25% of highly sensitized patients experience Antibody Mediated Rejection post-transplant and 85% of these Antibody Mediated Rejection episodes occur in the 1st post-transplant month, we feel the assessment of the potential impact of C1 INH therapy is best assessed in this time period. After completion of the C1 INH therapy, patients will be followed for an additional 6 month to assess allograft function and Antibody Mediated Rejection episodes as well as Donor Specific Antibodies.

The subjects will be followed to determine the proportion who develop evidence of Antibody Mediated Rejection within 6 month of completion of the study. In addition we will asses the transplanted patients to determine the number who sustain a viable and functioning kidney allograft for 6 months. All subjects will be evaluated on an intent-to-treat basis. The subject accrual rate will be limited to no more than five subjects per month in the initial three months to assure safety to all subjects. Repeat laboratories will be performed at the completion of C1 INH therapy to determine effect on levels and correlation with any potential events.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease.
* No known contraindications for therapy with Immune Globuillin Intravenous 10%/Rituximab or C1 INH.
* Age 18-65 years at the time of screening.
* Panel Reactive Antibody [PRA] > 50% demonstrated on 3 consecutive samples, Patient highly-HLA (Human Leukocyte Antigen) sensitized and a candidate for Living Donor/Deceased Donor transplantation after desensitization at Cedars Sinai Medical Center.
* At transplant, patient must have Donor Specific Antibody /Cross match + non-HLA (Human Leukocyte Antigen) identical donor.

Subject/Parent/Guardian must be able to understand and provide informed consent.

Exclusion Criteria:

* Lactating or pregnant females.
* Women of child-bearing age who are not willing or able to practice Food and Drug Administration [FDA]-approved forms of contraception.
* HIV-positive subjects.
* Subjects who test positive for Hepatitis B Virus infection [positive Hepatitis B Virus surface Antigen, Hepatitis B Virus core Antigen, or Hepatitis B Virus e Antigen/DNA] or Hepatitis C Virus infection [positive Anti-Hepatitis C Virus (EIA) and confirmatory Hepatitis C Virus Recombinant ImmunoBlot Assay (RIBA)].
* Subjects with active Tuberculosis.
* Subjects with selective Immunoglobulin A deficiency, those who have known anti-Immunoglobulin A antibodies, and those with a history of anaphylaxis or severe systemic responses to any part of the clinical trial material.
* Subjects who have received or for whom multiple organ transplants are planned.
* Recent recipients of any licensed or investigational live attenuated vaccine(s) within two months of the screening visit (including but not limited to any of the following:
* Adenovirus [Adenovirus vaccine live oral type 7] Varicella [Varivax] Hepatitis A [VAQTA] Rotavirus [Rotashield] Yellow fever [Y-F-Vax] Measles and mumps [Measles and mumps virus vaccine live] Measles, mumps, and rubella vaccine [M-M-R-II] Sabin oral polio vaccine Rabies vaccines [IMOVAX Rabies I.D., RabAvert])
* A significantly abnormal general serum screening lab result defined as a White Blood Cell < .0 X 103/ml, a Hemoglobin < 8.0 g/dL, a platelet count < 100 X 103/ml, , an Serum Glutamic Oxaloacetic Transaminase [SGOT] > 5X upper limit of normal, and an Serum Glutamic Pyruvic Transaminase [SGPT] >5X upper limit of normal range.
* Individuals deemed unable to comply with the protocol.
* Subjects with active Cytomegalovirus or Epstein Barr Virus infection as defined by Cytomegalovirus-specific serology (Immunoglobulin G or Immunoglobulin M) and confirmed by quantitative Polymerase Chain Reaction with or without a compatible illness.
* Subjects with a known history of previous myocardial infarction within one year of screening.
* Subjects with a history of clinically significant thrombotic episodes, and subjects with active peripheral vascular disease.
* Use of investigational agents within 4 weeks of participation.
* Know allergy/sensitivity to C1 INH infusions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley C Jordan, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai medical center, Los Angeles, California, United States

REFERENCES:
- [Background] Vo AA, Lukovsky M, Toyoda M, Wang J, Reinsmoen NL, Lai CH, Peng A, Villicana R, Jordan SC. Rituximab and intravenous immune globulin for desensitization during renal transplantation. N Engl J Med. 2008 Jul 17;359(3):242-51. doi: 10.1056/NEJMoa0707894. PMID 18635429
- [Background] Jordan SC, Tyan D, Stablein D, McIntosh M, Rose S, Vo A, Toyoda M, Davis C, Shapiro R, Adey D, Milliner D, Graff R, Steiner R, Ciancio G, Sahney S, Light J. Evaluation of intravenous immunoglobulin as an agent to lower allosensitization and improve transplantation in highly sensitized adult patients with end-stage renal disease: report of the NIH IG02 trial. J Am Soc Nephrol. 2004 Dec;15(12):3256-62. doi: 10.1097/01.ASN.0000145878.92906.9F. PMID 15579530
- [Background] Jordan SC, Reinsmoen N, Peng A, Lai CH, Cao K, Villicana R, Toyoda M, Kahwaji J, Vo AA. Advances in diagnosing and managing antibody-mediated rejection. Pediatr Nephrol. 2010 Oct;25(10):2035-45; quiz 2045-8. doi: 10.1007/s00467-009-1386-4. Epub 2010 Jan 14. PMID 20077121
- [Background] Solez K, Colvin RB, Racusen LC, Sis B, Halloran PF, Birk PE, Campbell PM, Cascalho M, Collins AB, Demetris AJ, Drachenberg CB, Gibson IW, Grimm PC, Haas M, Lerut E, Liapis H, Mannon RB, Marcus PB, Mengel M, Mihatsch MJ, Nankivell BJ, Nickeleit V, Papadimitriou JC, Platt JL, Randhawa P, Roberts I, Salinas-Madriga L, Salomon DR, Seron D, Sheaff M, Weening JJ. Banff '05 Meeting Report: differential diagnosis of chronic allograft injury and elimination of chronic allograft nephropathy ('CAN'). Am J Transplant. 2007 Mar;7(3):518-26. doi: 10.1111/j.1600-6143.2006.01688.x. PMID 17352710
- [Background] Shapiro R. Reducing antibody levels in patients undergoing transplantation. N Engl J Med. 2008 Jul 17;359(3):305-6. doi: 10.1056/NEJMe0804275. No abstract available. PMID 18635436
- [Result] Vo AA, Zeevi A, Choi J, Cisneros K, Toyoda M, Kahwaji J, Peng A, Villicana R, Puliyanda D, Reinsmoen N, Haas M, Jordan SC. A phase I/II placebo-controlled trial of C1-inhibitor for prevention of antibody-mediated rejection in HLA sensitized patients. Transplantation. 2015 Feb;99(2):299-308. doi: 10.1097/TP.0000000000000592. PMID 25606785

RESULTS

PARTICIPANT FLOW:
Groups:
- C1 Esterase Inhibitor: Patients receiving transplants will have pre-transplant labs for C1 INH levels, Complement 3 and Complement 4 obtained. In addition to the standard post-transplant immunosuppressive protocol, participating patients will receive 20 Units/kg C1 INH vs placebo (0.9% Normal Saline) on day 0 and day 2, then twice weekly X 3 weeks. A protocol biopsy will be performed at 6 month to assess the allograft for evidence of Antibody Mediated Rejection, including C4d staining using Banff 2009 criteria. After completion of the C1 INH therapy, patients will be followed up to 6M to assess allograft function and Anibody Mediated Rejection episodes as well as Donor Specific Antibody. A protocol biopsy will be performed at 6 month.
- Placebo: Patients will receive placebo (0.9% Normal Saline) on days 0 and day 2, then twice weekly for 3 weeks.
Period: Overall Study
Arm/Group | C1 Esterase Inhibitor | Placebo
Started | 10 (Transplant Day; Infusion #1 C1 esterase inhibitor vs Placebo) | 10 (Transplant Day; Infusion #1 C1 esterase inhibitor vs Placebo)
Day 2 | 10 (Infusion #2 C1 esterase inhibitor vs Placebo) | 10 (Infusion #2 C1 esterase inhibitor vs Placebo)
Week 2 | 10 (Infusion #3 C1 esterase inhibitor vs Placebo) | 10 (Infusion #3 C1 esterase inhibitor vs Placebo)
Week 2 | 10 (Infusion #4 C1 esterase inhibitor vs Placebo) | 10 (Infusion #4 C1 esterase inhibitor vs Placebo)
Week 3 | 10 (Infusion #5 C1 esterase inhibitor vs Placebo) | 10 (Infusion #5 C1 esterase inhibitor vs Placebo)
Week 3 | 10 (Infusion #6 C1 esterase inhibitor vs Placebo) | 10 (Infusion #6 C1 esterase inhibitor vs Placebo)
Week 4 | 10 (Infusion #7 C1 esterase inhibitor vs Placebo) | 10 (Infusion #7 C1 esterase inhibitor vs Placebo)
Week 4 | 10 (Infusion #8 C1 esterase inhibitor vs Placebo) | 10 (Infusion #8 C1 esterase inhibitor vs Placebo)
Month 1 | 10 | 10
Month 3 | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- C1 Esterase Inhibitor: Potential subjects will be identified after a review of medical records of patients under the care of one or more of the study investigators. Potential subjects will be identified and approached during an inpatient or outpatient clinical visit by a member of the research team. The Principal investigator (PI) I will explain what it means to be highly-sensitized and the risks associated with it. The PI will describe the study and explain the risks and benefits of participation. After the discussion, a copy of the consent form will be emailed or faxed to the patient for review & consideration of study participation. The patient can contact the study team to ask questions and sign the Informed Consent Form (ICF), if interested.
  C1 INH is dosed at 20 units per kg body weight and is administered by slow IV injection at a rate of approximately 4 mL per minute. Study patients will receive 20U/kg C1 INH vs placebo (0.9% NS) on days 0 and day 2, then twice weekly X 3 weeks.
- Placebo: Potential subjects will be identified after a review of medical records of patients under the care of one or more of the study investigators. Potential subjects will be identified and approached during an inpatient or outpatient clinical visit by a member of the research team. The Principal investigator (PI) I will explain what it means to be highly-sensitized and the risks associated with it. Then PI will describe the standard of care of Transplant Immunology Program (TIP) patients. After that PI will describe the study and explain the risks and benefits of participation. After the discussion, a copy of the consent form will be either emailed or faxed to the patient for review and consideration of study participation. The patient can contact the study team where they will have the opportunity to ask questions and then sign the Informed Consent Form (ICF), if interested.
- Total: Total of all reporting groups
Arm/Group | C1 Esterase Inhibitor | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (14) | 47 (16) | 47 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 2 | 7 | 9
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Post-transplant Biopsy to Identify Rejection Episodes
Description: Subjects will have a routine kidney biopsy 6 month after transplant to screen for episodes of acute rejection.
  For purposes of this investigation, antibody-mediated rejection (AMR) is defined as follows:
  * Deterioration of allograft function in a high-risk transplant recipient (i.e. sensitized patient with history of Donor Specific Antibodies) measured by serum Creatinine and estimated Glomerular Filtration Rate
  * Association with the presence of Donor Specific Antibody (usually increasing in strength) measured by luminex techniques.
  * Biopsy evidence of capillaritis, inflammation and C4d deposition.
Time Frame: 6 month
Population: 9 patients in each arm completed 6 month protocol biopsy. 1 patient in the placebo arm was withdrawn before 6M biopsy. 1 patient in treatment arm refused protocol biopsy.
Measure: Number; unit: Episode of rejection
Groups:
- C1 Esterase Inhibitor: 10 subjects will receive C1 esterase inhibitor in addition to standard of care immunosuppressive therapy.
  C1 Esterase Inhibitor: C1 Esterase Inhibitor 20 units/kg vs Placebo twice weekly x 4 weeks
- Normal Saline: 10 subjects placebo in addition to standard of care immunosuppressive therapy.
  C1 Esterase Inhibitor: C1 Esterase Inhibitor 20 units/kg vs Placebo twice weekly x 4 weeks
Arm/Group | C1 Esterase Inhibitor | Normal Saline
Number analyzed (Participants) | 9 | 9
Episode of rejection | 2 | 3

2. Secondary Outcome: Serum Creatinine
Description: Serum creatinine will be checked 6 months post transplant to monitor allograft function.
Time Frame: 6 months
Population: Mean serum creatinine levels at 6 month post-transplant from 10 patients in the C1 Esterase Inhibitor group and 10 patients in the placebo group were calculated.
Measure: Mean (Standard Deviation); unit: mg/dl (serum cr at 6m post transplant)
Groups:
- C1 Esterase Inhibitor: Patients receiving transplants will have pre-transplant labs for C1 INH levels, C3 and C4 obtained. In addition to the standard post-transplant immunosuppressive protocol, participating patients will receive 20 units/kg C1 INH vs placebo (0.9% NS) on day 0 and day 2, then twice weekly X 3 weeks (see Appendix A). A protocol biopsy will be performed at 6M to assess the allograft for evidence of AMR, including C4d staining using Banff 2009 criteria. After completion of the C1 INH therapy, patients will be followed up to 6M to assess allograft function and AMR episodes as well as DSA. A protocol biopsy will be performed at 6M.
- Placebo: Patients will receive placebo (0.9% NS) on days 0 and day 2, then twice weekly X3 weeks.
Arm/Group | C1 Esterase Inhibitor | Placebo
Number analyzed (Participants) | 10 | 10
mg/dl (serum cr at 6m post transplant) | 1.07 (0.39) | 1.08 (0.28)

3. Secondary Outcome: Donor Specific Antibodies [DSA] Class I
Description: Donor Specific Antibodies [DSAs] Class I will be checked 1, 3, and 6 months post transplant to monitor allograft function.
  DSA will be measured using a relative intensity score (RIS) ranges from 0 points = No DSA; 2 points = <5000MFI (weak intensity); 5 points = 5000-10,000 MFI (moderate intensty); 10 points = >10,000MFI (strong intensity). Each DSA can have a score of 10 maximum. However, patients may have more than one DSA and points can add up to more than 10. this depends on how many DSAs [Class I and/or Class II] are present at the time of transplant and quarterly after transplant. Patients can have an infinite number of donor specific antibodies, this score can be higher than 10.
Time Frame: 6 months
Population: Mean Donor Specific Antibody Class I levels at 1, 3, and 6 month post-transplant from 10 patients in the C1 Esterase Inhibitor group and 10 patients in the placebo group were calculated.
Measure: Mean (Standard Deviation); unit: DSA relative intensity score
Arm/Group | C1 Esterase Inhibitor | Placebo
Number analyzed (Participants) | 10 | 10
DSA relative intensity score | 10 (9.3) | 7.1 (4.8)

4. Secondary Outcome: Donor Specific Antibodies [DSA] Class II
Description: Donor Specific Antibodies [DSAs] Class I will be checked 1, 3, and 6 months post transplant to monitor allograft function.
  DSA will be measured using a relative intensity score (RIS) ranges from 0 points = No DSA; 2 points = <5000MFI (weak intensity); 5 points = 5000-10,000 MFI (moderate intensty); 10 points = >10,000MFI (strong intensity). Each DSA can have a score of 10 maximum. However, patients may have more than one DSA and points can add up to more than 10. this depends on how many DSAs [Class I and/or Class II] are present at the time of transplant and quarterly after transplant.
  However, patients may have more than one DSA and points can add up to more than 10 this depends on how many DSAs [Class I and/or Class II] are present at the time of transplant and quarterly after transplant. Patients can have an infinite number of donor specific antibodies, this score can be higher than 10.
Time Frame: 6 months
Population: Mean Donor Specific Antibody (DSA) Class II levels at 1, 3, and 6 month post-transplant from 10 patients in the C1 Esterase Inhibitor group and 10 patients in the placebo group were calculated.
Measure: Mean (Standard Deviation); unit: DSA relative intensity score
Arm/Group | C1 Esterase Inhibitor | Placebo
Number analyzed (Participants) | 10 | 10
DSA relative intensity score | 5.4 (3.2) | 9.0 (8.0)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Placebo: Total of 2 Serious Adverse Events (2/10 patients = 20%)
- C1 Esterase Inhibitor: Total of 1 Serious Adverse Event (1/10 = 10%)
Arm/Group | Placebo | C1 Esterase Inhibitor
Serious Adverse Events (participants affected / at risk) | 2/10 | 1/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=10) | C1 Esterase Inhibitor (N=10)
Post op Vascularization (Surgical and medical procedures) | 1/2 (1) | 0 (0) — Not related to study drug. Post op complication.
Hyperkalemia (Renal and urinary disorders) | 1 (1) | 0 (0) — Patient admitted post kidney transplant.
Perinephric Hematoma (Surgical and medical procedures) | 0 (0) | 1 (1) — Not related to study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No